CLINICAL TRIAL: NCT02211157
Title: Safety, Pharmacokinetics and Pharmacodynamics of BIRB 796 BS Tablets (20, 30, 150, 300, and 600 mg) Administered Orally to Healthy Human Subjects Once Daily for 7 Days. A Placebo Controlled, Randomised, Double Blinded Study
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BIRB 796 BS Tablets Administered to Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.3
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (3):
- BIBR 796 BS, fasted (Experimental): dose escalation
  Interventions: Drug: BIBR 796 BS
- BIBR 796 BS, fed (Experimental): 50 mg BIRB 796 BS (food effect)
  Interventions: Drug: BIBR 796 BS; Other: high fat breakfast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBR 796 BS
  Arms: BIBR 796 BS, fasted; BIBR 796 BS, fed
Drug: Placebo
  Arms: Placebo
Other: high fat breakfast
  Arms: BIBR 796 BS, fed

SUMMARY:
Study to assess safety, pharmacokinetics and pharmacodynamics of BIRB 796 BS in escalating multiple doses with and without a 64 g fat breakfast at the 50 mg dose level

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice and local legislation
* Age ≥ 18 and ≤ 45 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation > 400 ml within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the reference range of clinical relevance including, but not limited to total white cell count ≥ 10 x 10**9/L, C-reactive protein ≥ 4.5 mg/L, Gamma-Glutamyl Transferase ≥ 40 U/L, any hemoglobin or > 15 mg/dl protein or urine dipstick, abnormal Multitest® assessment of cellular immunity
* History of any familial bleeding disorder
* Inability to comply with dietary regimen of study centre

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2000-03; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant changes in laboratory parameters | up to day 16
Number of patients with abnormal findings in electrocardiogram (ECG) | up to day 16
Number of patients with adverse events | up to 30 days
Assessment of tolerability on a 4-point scale | day 16
Number of patients with clinically relevant changes in vital signs | up to 16 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for several time points | up to day 9
Area under the plasma concentration-time curve (AUC) for several time points | up to day 9
Time to maximum concentration (tmax) | up to day 9
Elimination rate constant (λz) | up to day 9
Terminal half-life (t1/2) | up to day 9
Mean residence time (MRT) | up to day 9
Apparent clearance (CL/f) | up to day 9
Apparent volume of distribution (Vz/F) | up to day 9
Assessment of neutrophil and monocyte activation by ex vivo stimulation of whole blood with formyl-methionyl-leucyl-phenylalanine (fMLP) | up to day 9
  Change in the Mac-1 / L-selectin ratio
Assessment of neutrophil and monocyte activation by ex vivo stimulation of whole blood with tumour necrosis factor (TNF) α | up to day 9
  Change in the Mac-1 / L-selectin ratio
Assessment of TNFα production by ex vivo stimulation of whole blood with endotoxin | up to day 9
Changes in cellular immune response measured by Multitest® | Day 8